CLINICAL TRIAL: NCT04202042
Title: Post-traumatic Stress Injuries Among Paramedics and Emergency Dispatchers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other)
Responsible Party: Principal Investigator, Steve Geoffrion, Researcher and Assistant professor, Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 162535
Record Dates: First submitted 2019-07-11; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Stress Disorders, Post-Traumatic; Acute Stress Disorder; Anxiety Disorders; Depressive Disorder; Substance Abuse; Absenteeism
Keywords: PFA; PTSD; Public safety personnel
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute; Anxiety Disorders; Depressive Disorder; Substance-Related Disorders | interventions — Psychological First Aid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological first aid (Experimental): PFA responders are trained to deliver 8 core actions in the aftermath of traumatic event (: contact and engagement, safety and comfort, stabilization, information gathering, practical assistance, connection with social supports, information on coping, and linkage with collaborative services (within the first 24 hours)
  Interventions: Other: Psychological first aid
- Usual organisational intervention (Active Comparator): One phone call by workplace psychologist (within the first 48 hours) and reference to employee aid program
  Interventions: Other: Usual organisational intervention

INTERVENTIONS:
Other: Psychological first aid — PFA responders (peer support workers) are trained to deliver 8 core actions: contact and engagement, safety and comfort, stabilization, information gathering, practical assistance, connection with social supports, information on coping, and linkage with collaborative services
  Arms: Psychological first aid
Other: Usual organisational intervention — Emergency intervention by workplace psychologist and limited therapeutic sessions with employee aid program
  Arms: Usual organisational intervention

SUMMARY:
As part of their work, emergency first responders, such as paramedics and emergency medical dispatchers are exposed daily to traumatic events. These traumatic events can have many impacts on mental health, such as acute stress disorder and post-traumatic stress disorder. Research has shown that intervening early after exposure to a traumatic event helps to identify people at risk and to prevent post-traumatic stress disorder. The Psychological First Aid approach originally developed for mass traumas, is an intervention advocated by international experts today following a traumatic event. However, this approach is still very little studied, especially when it is part of an organization of emergency first responders. It therefore still lacks scientific validity. The main objective of this research will be to assess whether the Psychological First Aid program provided by peer-support workers helps to reduce the initial distress caused by traumatic events and to foster short- and long-term adaptive functioning and coping.

DETAILED DESCRIPTION:
In May 2018, Urgences-Santé (i.e., EMT corporation for the Montreal area) implemented PFA as a peer-support intervention for EMT affected by traumatic events in the course of their work. In collaboration with Urgences-Santé, this project aims to evaluate the feasibility of PFA as a post-traumatic peer-support intervention among EMT. Feasibility studies are used to determine whether an intervention should be recommended for efficacy testing when there are few previously published studies or existing data using a specific intervention technique. This catalyst project relies on participatory research principles. With Urgences-Santé stakeholders, three specific research objectives were elaborated in order to answer the question "Can PFA work for EMT?":

1. To assess the acceptability of PFA for EMT;
2. To assess the implementation of PFA in Urgences-Santé;
3. To test the limited-efficacy (i.e., efficacy within limitations such as small sample size and convenience sampling of PFA among Urgences-Santé trauma-exposed EMT).

Based on the few studies that assess different aspects of the feasibility of PFA in high-risk organizations, this project relies on three working hypotheses. First, we expect that PFA be acceptable among EMT. Second, we stipulate that few obstacles limited the implementation of PFA in Urgences-Santé given that this organization followed Forbes' implementation framework and favored a train-the-trainer approach. Third, we foresee that PFA will accelerate the recovery process of EMT, as measured by a greater decrease in PTSI, heart rate and absenteeism in the days following the traumatic event among those who received PFA compared to those who received the standard intervention (i.e., reference to employee aid program). If confirmed, these hypotheses will allow us to affirm that PFA can work as a post-traumatic intervention among EMT for the prevention of PTSI. Our results would therefore represent a catalyst towards a larger RCT that would answer the question "Does PFA work for EMT?" with an adequate sample size.

ELIGIBILITY:
Inclusion Criteria:

* Actively working at Urgence-Santé organization as paramedics or emergency medical dispatchers
* Exposed to a traumatic event at work (after the baseline)

Exclusion Criteria:

- at high risk of suicidal behaviour

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Change in acute stress symptoms | 2 times after exposure to the traumatic event; 48-72 hours (T1), 7 to 9 days (T2)
  The Acute Stress Disorder Scale (Bryant, Moulds et Guthrie, 2000) Scores : 1 to 5, higher scores mean worse outcome.
Change in post-traumatic stress symptoms | Baseline (T0) + 2 times after exposure to the traumatic event; 30 to 32 days (T3), 90 to 95 days (T4)
  The Post-Traumatic Checklist-5 (Ashbaugh, Houle-Johnson, Herbert, El-Hage et Brunet, 2016) Scores : 0 to 4, higher scores mean worse outcome.
Change in depressive symptoms | 4 times after exposure to the traumatic event; 48-72 hours (T1), 7 to 9 days (T2), 30 to 32 days (T3), 90 to 95 days (T4)
  The Patient Health Questionnaire-9 (Kroenke, Spitzer & Williams, 2001) Scores : 0 to 3, higher scores mean worse outcome.
Change in anxiety symptoms | 4 times after exposure to the traumatic event; 48-72 hours (T1), 7 to 9 days (T2), 30 to 32 days (T3), 90 to 95 days (T4)
  The General Anxiety Disorder-7 scale (Spitzer, Kroenke, Williams & Löwe, 2006) Scores : 0 to 3, higher scores mean worse outcome
Change in substance abuse : alcohol | 4 times after exposure to the traumatic event; 48-72 hours (T1), 7 to 9 days (T2), 30 to 32 days (T3), 90 to 95 days (T4)
  The Alcohol Use Disorders Identification Test (Saunders, Aasland, Babor, de la Fuente & Grant, 1993) Scores : 0 to 5, higher scores mean worse outcome
Change in substance abuse : drug | 4 times after exposure to the traumatic event; 48-72 hours (T1), 7 to 9 days (T2), 30 to 32 days (T3), 90 to 95 days (T4)
  The Drug Abuse Screening Test (Villalobos-Gallegos, Perez-Lopez, Graue-Moreno, Marin-Navarrete & Mendoza-Hassey, 2015) Scores : Yes or No, higher "Yes" answers mean worse outcome

SECONDARY OUTCOMES:
Change in heart rate variation | Baseline (T0) + each week until 90 to 95 days after the event
  Manual measurement (wrist or neck) of the resting heart rate at each measurement time Scores = pulse per minute, higher scores mean worse outcome
Absenteeism at work | 90 to 95 days after the traumatic event (T4)
  Number of days taken off of work for psychological reasons from the time of traumatic exposure up to T4. Information requested directly from participants in the questionnaire set.

CONTACTS AND LOCATIONS:
Overall Officials: Luc De Montigny, Principal Investigator — Urgences-santé; Stephane Guay, Principal Investigator — Research Center of the Institut universitaire en santé mentale de Montréal
Locations (1):
- Urgences-santé, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bryant RA. Acute stress reactions: can biological responses predict posttraumatic stress disorder? CNS Spectr. 2003 Sep;8(9):668-74. doi: 10.1017/s1092852900008853. PMID 15079140
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders DSM-5 (5e éd.). Arlington, VA: American Psychiatric Publishing
- [Background] Brymer, M. Jacobs, A. Layne, C., Pynoos, R., Ruzek, J., Steinberg, A., Vernberg. E. & Watson, P. (2006). Psychological First Aid: Field Operations Guide: 2nd Edition. National Child Traumatic Stress Network. Doi:10.1037/e536202011-001
- [Background] Ruzek, J. I., Brymer, M. J., Jacobs, A. K., Layne, C. M., Vernberg, E. M. & Watson, P. J. (2007). Psychological first aid. Journal of Mental Health Counseling, 29(1), 17-49.
- [Background] Guidelines for the Management of Conditions Specifically Related to Stress. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK159725/ PMID 24049868
- [Background] Bryant RA, Moulds ML, Guthrie RM. Acute Stress Disorder Scale: a self-report measure of acute stress disorder. Psychol Assess. 2000 Mar;12(1):61-8. PMID 10752364
- [Background] Ashbaugh AR, Houle-Johnson S, Herbert C, El-Hage W, Brunet A. Psychometric Validation of the English and French Versions of the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). PLoS One. 2016 Oct 10;11(10):e0161645. doi: 10.1371/journal.pone.0161645. eCollection 2016. PMID 27723815
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Villalobos-Gallegos, L., Perez-Lopez, A., Graue-Moreno, J., Marin-Navarrete, R., & Mendoza-Hassey, R. (2015). Psychometric and diagnostic properties of the Drug Abuse Screening Test (DAST): Comparing the DAST-20 vs. the DAST-10. Salud Mental, 38, 2, 89-94.
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902